CLINICAL TRIAL: NCT01193231
Title: A Single Center, Randomized, Contralateral, 6 Month Study to Evaluate the Safety, Analgesic Efficacy of ACUVAIL™ (Ketorolac Tromethamine Ophthalmic Solution) 0.45%, in Post-PRK Corneal Wound Healing
Brief Title: A 6 Month Study to Evaluate the Safety, Analgesic Efficacy of ACUVAIL™ (Ketorolac Tromethamine Ophthalmic Solution) 0.45%, in Post-PRK Corneal Wound Healing
Status: Completed | Type: Observational
Sponsor: Durrie Vision (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Daniel S. Durrie, MD, Presidenet, Durrie Vision
Other Study IDs: ACVL-001
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Must be PRK Candidate
Keywords: Laser Vision Correction; Photorefractive Keratectomy; PRK; Nearsighted; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acuvail 0.45%: Each subject will be randomized to the eye that they will use Acuvail in for 3 days after PRK
- Systane Ultra Preservative Free Tears: Each subject's contralateral eye (other eye) will use Sytane for 3 days after PRK surgery.

SUMMARY:
STUDY OBJECTIVE: To evaluate the safety and efficacy of Acuvail 0.45% administered BID for increasing corneal re-epithelialization, decreasing the time to zero pain in post-photorefractive keratectomy (PRK) surgery, and PRK enhancement assessment at 6 months post op

CLINICAL HYPOTHESES: Acuvail 0.45% administered twice daily is superior to Systane Ultra lubricant in treating post PRK pain

OVERAL STUDY DESIGN:

Structure: Single-center, randomized, open label, contralateral (one eye receives Acuvail, one eye Systane Ultra)

Treatment Group: Patients will be randomized to the eye that will receive Acuvail 0.45% Assignment: Acuvail 0.45% in one eye, Systane Ultra in contralateral eye

Duration: 6.5 months

Controls: Systane Ultra preservative-free lubricant

Dosage/Dose Regimen: Study medication will be administered to the randomized eye through post op days 1-2 BID

Visit Schedule: Screening (baseline), Day 2-30 (Surgery), post surgery Day 1 and each day through corneal re-epithelialization, post surgery months 1, 3, and 6.

Number of Patients: 10 (20 eyes)

Condition/Disease: patients undergoing bilateral PRK surgery

DETAILED DESCRIPTION:
1. INTRODUCTION

   Laser Vision Correction is one of the most commonly performed elective procedures in the United States. Although the Laser in situ keratomileusis (LASIK) is the more popular vision correction procedure, a growing number of surgeons have switched to surface ablation techniques, including PRK, LASEK, and Epi-LASIK. In surface laser procedures, the epithelium (clear outer skin of the cornea) is removed, prior to laser reshaping of the cornea. This creates an epithelial defect that can take 3-6 days for the epithelium to regenerate. During this healing process, patients often report moderate to severe ocular pain.

   A variety of treatments have been utilized to reduce postoperative pain. Placement of a contact lens on the eye immediate post PRK, has been shown to reduce patient discomfort as well as topical dilute tetracaine, oral medications, and even prednisone has been recommended as treatment options for pain control. Another method that has been shown in a number of studies to assist with the reduction of post operative pain is topical non steroidal anti inflammatory drops.

   Pain management following PRK surgery has been minimized by more advanced surgical techniques, antibiotics, and pre- or post-operative use of topical NSAID solutions. We will compare the use of Acuvail 0.45% administered twice daily to Systane Ultra in treating post PRK pain.
2. STUDY OBJECTIVE

   To evaluate the safety and efficacy of Acuvail 0.45% administered BID for increasing re-epithelialization time, decreasing the time to zero pain in post-photorefractive keratectomy (PRK) surgery and assessment of PRK enhancement needs at 6 months post op.

   CLINICAL HYPOTHESES: Acuvail 0.45% administered twice daily is superior to Systane Ultra in treating post PRK pain

   Efficacy Objectives

   Primary: Time to re-epithelialization Secondary: Time to zero pain as documented in Patient Comfort Questionnaire PRK enhancement assessment at 6 month post op

   Safety Measures: Visual recovery-UCVA & BCVA IOP Biomicroscopy Adverse Events Optovue OCT-epithelial image Pachymetry Pregnancy test
3. STUDY DESIGN

This is a Phase 4, single-center, open label, randomized, contralateral (one eye receives Acuvail, one eye Systane Ultra Lubricant Eye Drops). Patients will be randomized to the eye that will receive Acuvail 0.45%. The duration of the study is estimated to be approximately 6.5 months for each study subject enrolled.

Controls: Systane Ultra preservative free tears

Dosage/Dose Regimen: Study medication will be administered twice a day to the randomized eye days 1-3 post operatively BID

Visit Schedule: Screening (baseline), Day 2-30 (Surgery), post surgery Day 1, Day 2, Day 3, and each day through corneal re-epithelialization, post surgery months 1, 3, and 6.

Number of Patients: 10- all subjects will use study medication in one eye, and Systane Ultra in the other eye

Condition/Disease: patients undergoing bilateral PRK surgery

Instructions for storage, use and administration Study medication and control medication should be stored in a secure area at room temperature and administered to patients entered in to the study in accordance to this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 18-39 yrs of age, in good general health
2. Patient is schedule to undergo bilateral PRK surgery
3. The difference between the two eyes ≤ 2 D
4. Refractive error -1 to -8 diopters (spherical equivalent) at baseline
5. Females of childbearing potiential must have a negative pregnancy test result at baseline. A female considered to be of non-childbearing potential is she is postmenopausal (no menses for 12 consecutive months) or is without a uterus.
6. Ability to follow study instructions and likely to complete the entire course of the study
7. Written informed consent has been obtained
8. Written HIPPA authorization has been obtained

Exclusion Criteria:

1. Uncontrolled systemic disease
2. Any active ocular disease, corneal abnormalities, lid abnormalities, or any ocular pathologies
3. History of serious eye disease, trauma, or previous ocular surgery
4. History of unstable myopia
5. History of herpes keratitis
6. Known allergy or hypersensitivity to the study medication
7. Anticipated wearing of contact lenses in addition to the required bandage contact lens post-PRK. Patients who wear soft contact lenses should discontinue wearing them at least 3 days prior to baseline visit. Patients wearing RGP or hard contact lenses should discontinue wearing them at least 3 weeks prior to baseline visit.
8. Females who are pregnant, breastfeeding, or trying to conceive.
9. Keratoconus or keratoconus suspect
10. Concurrent participation in an investigational drug study or participation within 30 days prior to study start
11. Any condition or situation which, in the investigator's opinion, may put patient at significant risk or may confound the study results

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male or female patients, 18-39 yrs of age, in good general health Patient is schedule to undergo bilateral PRK surgery The difference between the two eyes ≤ 2 D Refractive error -1 to -8 diopters (spherical equivalent) at baseline
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time to re-epithelialization | 3-7 days
  Amount of days it takes for the cornea to re-epithelialize after PRK surgery, will be documented for each eye separately.

SECONDARY OUTCOMES:
Time to zero pain | 3-7 days
  Study subject will complete a questionnaire about their comfort levels at each postoperative visit, up to an including the 6 month post op exam.
Occurence of enhancments | 6 months post operative
  Will document the number of requested/recommended enhancement procedures at the 6 month postoperativ visit.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Durrie, MD, Principal Investigator — Durrie Vision
Locations (1):
- Durrie Vision, Overland Park, Kansas, United States